CLINICAL TRIAL: NCT05635474
Title: Effects of Bacillus Coagulans TCI711 Supplementation on Liver and Gut Microbiota Function in Non-alcoholic Fatty Liver Disease Patients
Brief Title: Effects of Bacillus Coagulans on Liver and Gut Microbiota Function in NAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Collaborators: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: N202208021
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Effects of Bacillus Coagulans TCI711 Supplementation on Liver and Gut Microbiota Function in Non-alcoholic Fatty Liver Disease Patients
MeSH Terms: interventions — exopolysaccharide biopolymer, Bacillus coagulans

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dietary supplement (Experimental): According to the 2018 statistics of the American Association of Liver Diseases, about 25% of the world's population has non-alcoholic fatty liver disease. Bacillus coagulans does not exist in intestinal microbiota, because it has characteristics of spore production and lactobacillus lactic acid production, and has the ability to maintain the health of intestinal bacteria, acid and alkali resistance, With the advantages of high temperature resistance and high stability, it is currently one of the commonly used probiotic strains. Clinical studies have shown that after intervention of a single Bacillus coagulans strain in patients with non-alcoholic fatty liver disease, the problem of liver fat accumulation and inflammation can be significantly improved, so supplementing Bacillus coagulans TCI711 probiotics isolated from apples may improve Functions of liver and gut microbiota in patients with nonalcoholic fatty liver disease.
  Interventions: Dietary Supplement: Bacillus Coagulans
- placebo (Placebo Comparator): The placebo was also given in the form of capsules, the main ingredients were maltodextrin, silicon dioxide and magnesium stearate
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bacillus Coagulans — Bacillus coagulans is a Gram-positive bacterium belonging to the genus Bacillus and does not exist in the intestinal microbiota, because it has the characteristics of spore production and lactobacillus lactic acid production, and has the ability to maintain the health of intestinal bacteria, acid and alkali resistance, With the advantages of high temperature resistance and high stability, it is currently one of the commonly used probiotic strains.
  Arms: dietary supplement
Dietary Supplement: Placebo — The placebo was also administered in the form of capsules consisting of maltodextrin, silicon dioxide, and magnesium stearate.
  Arms: placebo

SUMMARY:
According to the 2018 statistics of the American Association of Liver Diseases, about 25% of the world's population has non-alcoholic fatty liver disease, and about 10 to 20% of patients with simple fatty liver will develop non-alcoholic steatohepatitis, and about 25 to 50% of non-alcoholic fatty liver patients will continue to develop liver fibrosis, which may even lead to liver cirrhosis or liver cancer, so how to improve the liver fat accumulation of non-alcoholic fatty liver patients is one of the topics that scholars in related fields have paid attention to in recent years . Bacillus coagulans is a Gram-positive bacterium belonging to the genus Bacillus and does not exist in the intestinal microbiota, because it has the characteristics of spore production and lactobacillus lactic acid production, and has the ability to maintain the health of intestinal bacteria, acid and alkali resistance, With the advantages of high temperature resistance and high stability, it is currently one of the commonly used probiotic strains. Clinical studies have shown that after intervention of a single Bacillus coagulans strain in patients with non-alcoholic fatty liver disease, the problem of liver fat accumulation and inflammation can be significantly improved, so supplementing Bacillus coagulans TCI711 probiotics isolated from apples may improve Functions of liver and gut microbiota in patients with nonalcoholic fatty liver disease. Therefore, this experiment is to investigate the effect of supplementing Bacillus coagulans TCI711 probiotics on the function of liver and intestinal flora in fatty liver patients.

DETAILED DESCRIPTION:
According to the 2018 statistics of the American Association of Liver Diseases, about 25% of the world's population has non-alcoholic fatty liver disease, and about 10 to 20% of patients with simple fatty liver will develop non-alcoholic steatohepatitis, and about 25 to 50% of non-alcoholic fatty liver patients will continue to develop liver fibrosis, which may even lead to liver cirrhosis or liver cancer, so how to improve the liver fat accumulation of non-alcoholic fatty liver patients is one of the topics that scholars in related fields have paid attention to in recent years . Bacillus coagulans is a Gram-positive bacterium belonging to the genus Bacillus and does not exist in the intestinal microbiota, because it has the characteristics of spore production and lactobacillus lactic acid production, and has the ability to maintain the health of intestinal bacteria, acid and alkali resistance, With the advantages of high temperature resistance and high stability, it is currently one of the commonly used probiotic strains. Clinical studies have shown that after intervention of a single Bacillus coagulans strain in patients with non-alcoholic fatty liver disease, the problem of liver fat accumulation and inflammation can be significantly improved, so supplementing Bacillus coagulans TCI711 probiotics isolated from apples may improve Functions of liver and gut microbiota in patients with nonalcoholic fatty liver disease. Therefore, this experiment is to investigate the effect of supplementing Bacillus coagulans TCI711 probiotics on the function of liver and intestinal flora in fatty liver patients.

All the participants in the experiment were subjected to body position measurement, blood and feces collection, liver fiber analyzer analysis and questionnaire survey before supplementation. Afterwards, the subjects were divided into the experimental group and the placebo group in a random and double-blind manner. The experimental group was given Participants ingested one capsule containing the Bacillus coagulans TCI711 probiotic daily for 8 weeks, while the placebo group received a placebo-only capsule. All participants in the experiment took body position measurement and questionnaire survey again 4 weeks after supplementation, and body position measurement, blood and feces collection, liver fiber analyzer analysis and questionnaire survey again 12 weeks after supplementation. Blood was collected once each time, and 24 mL of blood was collected each time, and a total of 48 mL of blood was collected to evaluate the benefit of supplementing Bacillus coagulans TCI711 probiotics.

Bacillus coagulans TCI711 probiotics are expected to be beneficial to liver and intestinal flora functions in patients with fatty liver disease.

ELIGIBILITY:
Inclusion Criteria:

* 20-75 years old adult
* Have fatty liver disease

Exclusion Criteria:

* History of hepatitis B, hepatitis C, cirrhosis, liver fibrosis, or bariatric surgery
* Controlled attenuation parameter for fatty liver degeneration < 220 dB/m
* Have taken antibiotics within 3 months
* Have participated in any trial or research project within 3 months
* Taking any nutritional supplements during the trial
* Diet without maintaining daily habits and avoiding alcohol intake

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-25 (Actual); Primary Completion 2022-12-05 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Fibroscan | two month
  Liver fibrometer (Echosens, Paris, France) can be quantified with specific numerical values, which can be used at the same time The degree of fatty liver and liver fibrosis can be detected in real time by measuring LSM and CAP by transient elastography (Shrestha et al., 2021). During the measurement, the patient is in a supine position, the right arm is abducted, the forearm is under the head, and the right side of the body is bare and slightly raised. The physician uses the ultrasound gel-covered probe tip to place in the intercostal space above the right liver lobe, and uses A mode Image localization of liver sections that are at least 6 cm thick and free of any large vascular structures, and the probe button is pressed for image acquisition, which measures in the depth range of 25-45 mm (Shrestha et al., 2021).

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical university, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided